CLINICAL TRIAL: NCT05680467
Title: Short-term Effects of Manual Therapy Plus Capacitive and Resistive Electric Transfer Therapy in Pain Disability and Spinal Mobility in Individuals With Chronic Low Back Pain: A Randomized Clinical Trial Study
Brief Title: Manual Therapy Plus Capacitive and Resistive Electric Transfer Therapy in Individuals With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Hellenic University (Other)
Responsible Party: Principal Investigator, Dimitrios Lytras, Dimitrios Lytras, Principal Investigator, Senior Lecturer of Physiotherapy, International Hellenic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC-06/2022
Record Dates: First submitted 2022-12-24; First posted 2023-01-11 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Chronic Low Back Pain
Keywords: Chronic Low back pain; Manual therapy; Capacitive and Resistive Electric Transfer Therapy
MeSH Terms: interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: Sixty participants with chronic low back pain will be randomly assigned to three groups of 20 each. The allocation of the sample to the groups will be performed using a randomization program (https://www.randomizer.org/) by an independent researcher. In the first group, a manual protocol will be applied with the simultaneous application of a high-frequency current through TECAR, in the second group, the same manual protocol will be applied without the TECAR device, while the third group will not receive any treatment. Participants of the two intervention groups will follow a total of six treatments over a period of three weeks with a follow-up after one month.
Who Masked: Outcomes Assessor
Masking Description: A masked assessor will conduct the measurements
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- "Soft Tissue Mobilization" (Experimental): Participants allocated to this group will receive six sessions of soft tissue mobilization technique accord to Kaltenborn (2018) .
  Interventions: Other: Manual Therapy
- "Soft Tissue Mobilization" and "TECAR" (Experimental): Participants allocated to this group will receive the same manual therapy protocol with Group 1 in combination with Capacitive and Resistive Electric Transfer Therapy (TECAR).
  Interventions: Other: Manual Therapy plus TECAR
- "Control" (Active Comparator): Control Group
  Interventions: Other: Control

INTERVENTIONS:
Other: Manual Therapy — The protocol will last 30 minutes and will include the application of the following manual techniques:
  * Lumbar soft tissue and joint cranial and lateral mobilization with the patient in the supine position
  * Bilateral medial lumbar soft tissue mobilization
  * Functional massage on the quadratus lumborum muscle with the patient in a lateral position on both sides
  * Extension with coupled sidebending mobilization of the thoracic area with the patient in a lateral position on both sides
  * Soft tissue lateral mobilization of the thoracic area with the patient in a lateral position on both sides
  Arms: "Soft Tissue Mobilization"
Other: Manual Therapy plus TECAR — The participants of this group will be given the same manual protocol as the first group in combination with the application of high frequency current. Soft tissue mobilization manipulations will be applied in combination with a capacitive conventional electrode and with a special electrode bracelet that makes the therapist's own hand as an antistatic electrode. The frequencies of the high frequency current will be 300khz, 500khz, and 1MHz, while as a reference electrode a flexible self-adhesive ground will be used placed on the abdomen
  Arms: "Soft Tissue Mobilization" and "TECAR"
Other: Control — Participants in this group will only receive general instructions about managing their back pain and counseling about avoiding activities that may worsen their symptoms.
  Arms: "Control"

SUMMARY:
Chronic low back pain is defined as back pain that lasts longer than 12 weeks. The aim of this clinical study is to investigate the efficacy of combining a program of manual techniques with the application of Capacitive and Resistive Electric Transfer (TECAR) therapy to treat chronic low back pain. Sixty adults with chronic low back pain will be randomly divided into three groups of 20 each. In the participants of the first group, a therapeutic protocol of manual soft tissue mobilization in the lumbar region will be applied. To the participants of the second group, the same protocol of manual techniques will be applied in combination with TECAR therapy, which will be applied through a conventional capacitive electrode as well as an antistatic electrode bracelet (making the hand of the physical therapist an antistatic electrode). The third group participants will receive no treatment. Both programs will include six treatments over two weeks. Pain in the last 24 hours with the Numeric Pain Rating Scale (NPRS), functional ability with the Roland-Morris Disability Questionnaire (RMDQ), Pressure Pain Threshold (PPT) in the lumbar region with an algometer, and lumbar flexion range of motion through fingertip-to-floor distance (FFD) test will be evaluated before and after the intervention with a follow-up one month later. For the statistical analysis of the results, a two-factor analysis of variance with repeated measurements will be applied, while the statistical significance index will be set at p < .05.

DETAILED DESCRIPTION:
Background: Chronic low back pain is defined as back pain that lasts longer than 12 weeks.

Aim: The purpose of this clinical study is to investigate the efficacy of combining a program of manual techniques with the application of Capacitive and Resistive Electric Transfer (TECAR) therapy in people with chronic low back pain.

Method: Sixty adults with chronic low back pain will be randomly divided into three groups of 20 people each. In the participants of the first group, a therapeutic protocol of manual soft tissue mobilization in the lumbar region will be applied. To the participants of the second group, the same protocol of manual techniques will be applied in combination with TECAR therapy, which will be applied through a conventional capacitive electrode as well as an antistatic electrode bracelet (making the hand of the physical therapist an antistatic electrode). The third group participants will receive no treatment. Both programs will include six treatments over two weeks. Pain in the last 24 hours with the Numeric Pain Rating Scale (NPRS), functional ability with the Roland-Morris Disability Questionnaire (RMDQ), Pressure Pain Threshold (PPT) in the lumbar region with an algometer, and lumbar flexion range of motion through fingertip-to-floor distance (FFD) test will be evaluated before and after the intervention with a follow-up one month later. For the statistical analysis of the results, a two-factor analysis of variance with repeated measurements will be applied, while the statistical significance index will be set at p < .05.

Expected results: The protocol proposed in this clinical study combines the beneficial effects of TECAR treatment with the benefits of applying manual techniques. Modern TECAR devices make it possible, through special resistive bracelet electrodes, to turn the hand of the therapist into a mobile electrode providing a simultaneous effect of the two therapeutic means through manual techniques and high-frequency current. For this reason, we expect the specific combination to be more effective than the individual application of manual techniques in improving the clinical picture of adults with chronic low back pain. For the statistical analysis of the results, a two-way ANOVA with repeated measurements will be applied.

ELIGIBILITY:
Inclusion Criteria:

* Duration of symptoms 12 weeks
* Women - Men
* Age range between 20 and 60 years
* Written consent to participate in the study

Exclusion Criteria:

* Neuropathic pain extending along the lower limb due to nerve root compression
* Previous spine surgery
* History of spine trauma or fracture
* Implanted pacemakers
* Pregnancy
* Cancer
* Systemic musculoskeletal diseases, diagnosed neurodegenerative diseases (e.g., Parkinson's), epilepsy, and history of psychiatric disorders

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Changes in low back pain intensity with Numeric Pain Rating Scale (NPRS) | pre-treatment, week: 1, 2, 6
  This tool is an eleven-point pain scale numbered from zero to 10. The left end of the scale corresponds to zero and is marked as "No pain", whereas the right end corresponds to 10 and is marked as "Maximum pain". Consequently, a higher value indicates more intense pain (Childs et al, 2005). The examinee is asked to choose an integer that best reflects the intensity of their pain. The NPRS is widely used to measure pain in both clinical practice and research, showing high test-retest reliability and high conceptual construct validity.
Changes in Pressure Pain Threshold (PPT) with pressure algometry | pre-treatment, week: 1, 2, 6
  Pressure pain threshold (PPT) is defined as the minimal amount of pressure that produces pain. PPT will be assessed by a digital algometer and will be evaluated bilaterally in the quadratus lumborum muscle, in the sacroiliac joints, and paravertebrally in the L4-L5 intervertebral space. The metal rod of the algometer will be placed vertically on the site and the examiner will apply gradually increasing pressure at a rate of 1Kg/s. PPT is calculated in kg/cm2 (Imamura et al., 2016)
Changes in functional capacity with the Greek Version of Roland-Morris Disability Questionnaire (RMDQ) | pre-treatment, week: 1, 2, 6
  The functional ability of the participants will be evaluated with the Greek version of the Roland-Morris questionnaire, which consists of 24 questions related to daily activities that patients often report difficulty performing due to low back pain. Each positive answer earns one point and the final score is calculated by adding all the points. Therefore, the higher the score, the greater the restriction. The Greek version of the questionnaire shows satisfactory reliability and validity (ICC: 0.44-0.92) (Boscainos et al., 2003).
Changes in lumbar spine flexion range of motion with the Fingertip-To-Floor Test | Time Frame: pre-treatment, week: 1, 2, 6
  Range of trunk forward flexion will be assessed through the Fingertip-To-Floor Test. When performing the test, the examinee is asked to try to reach the ground with the fingers of their hands by leaning forward while keeping their knees and hips extended. The examiner measures with a tape the distance of the fingers from the ground. The test is widely used in clinical practice to measure spinal mobility and shows high reliability and validity indices (Ekedahl et al. 2010).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physiotherapy, Faculty of Health Sciences International Hellenic Universit, Thessaloniki, Sindos Thessaloníki, Greece

IPD SHARING:
Plan to Share IPD: No